CLINICAL TRIAL: NCT02786563
Title: Changes in Ultrasonographic Assessment of Inflammation Upon Initiation of Adalimumab Combination Therapy in Chinese Rheumatoid Arthritis Patients With Inadequate Response to Methotrexate
Brief Title: Changes in Ultrasonographic Assessment of Inflammation Upon Initiation of Adalimumab Combination Therapy in Chinese Rheumatoid Arthritis (RA) Patients With Inadequate Response to Methotrexate
Status: Withdrawn | Type: Observational
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-074
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: power doppler (PD); ultrasonographic (US); rheumatoid arthritis (RA); disease activity scale (DAS); C-reactive protein (CRP)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with RA receiving adalimumab: This group contains participants in China with RA receiving adalimumab

SUMMARY:
Prospective, post-marketing, multi-center, open-label study to explore if the initiation of adalimumab could influence grey-scale (GS) and power Doppler (PD) ultrasonographic (US) score using 36-joint plus 4-tendon scoring system, and validate the applicability of different simplified US joint scoring systems.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe RA despite treatment with methotrexate (MTX).
* Eligible to use adalimumab according to the local label without any contraindication.
* Naïve to adalimumab, and participants with prior exposure to any other biologic disease-modifying antirheumatic drugs (DMARDs) should have experienced at least five half-lives of the biologics after treatment discontinuation.
* Participants for whom investigators decided to prescribe adalimumab as per local label and are initiating adalimumab at baseline.

Exclusion Criteria:

* Other inflammatory condition which may affect the signs on joints ultrasound (eg, gouty arthritis, or other chronic rheumatic disease besides RA).
* Currently being treated with or has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days of the baseline visit.
* Participants with contraindication or are not appropriate to use adalimumab according to local label or investigators' judgment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving adalimumab with Rheumatoid Arthritis (RA) in China
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in grey-scale (GS) scores | Week 0 (baseline) and Week 12
  Change in GS scores from baseline at Week 12, using 36-joint scoring system
Change in power Doppler (PD) semi-quantitative scores from baseline | Week 0 (baseline) and Week 12
  Change in PD semi-quantitative scores from baseline at week 12, using 36-joint scoring system
Correlation between the 36-joint plus 4-tendon assessment versus simplified joint power Doppler (PD) ultrasonographic (US) assessments, which include 12-joint/7-joint/6-joint plus 4-tendon systems. | Week 0 (baseline) and Week 12
  Correlation coefficients will be presented to assess the correlation between the 36-joint plus 4-tendon PDUS assessment versus the simplified 12-joint/7-joint/6-joint plus 4-tendon assessments.

SECONDARY OUTCOMES:
Change from baseline in counts of joints with US detected bone erosion | Baseline (Week 0) to Week 12
  The change in counts of joints with US detected bone erosion.
Percentage of participants achieving low disease activity | Baseline (Week 0) to Week 12 and Week 20
  The percentage of participants achieving low disease activity (LDA, DAS 28-CRP greater than or equal to 2.6 but less than 3.2).
Correlation between changes of 36-joint plus 4-tendon PDUS score and disease activity DAS 28-CRP. | Baseline (Week 0) to Week 20
Percentage of patients achieving clinical remission | Baseline (Week 0) to Week 12 and Week 20
  The percentage of participants achieving clinical remission (DAS 28-CRP less than 2.6).
Change in DAS 28-CRP from baseline | Baseline (Week 0) to Week 12 and Week 20
  The Disease Activity Score C-Reactive Protein (DAS 28-CRP); 4 variables, using 28-joint counts and CRP.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (4):
- China (4):
  - Peking University Peoples Hospit /ID# 148961, Beijing, Beijing Municipality
  - Xijing Hospital /ID# 148960, Xi'an, Shaanxi
  - Hosp Ppl Liberation Army 301 /ID# 148962, Beijing
  - Renji Hosp, Shanghai Jiaotong /ID# 148959, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com/